CLINICAL TRIAL: NCT02039219
Title: A Double-Blind, Placebo-Controlled Trial of Obeticholic Acid in Patients With Moderately Severe Alcoholic Hepatitis (AH)
Brief Title: Trial of Obeticholic Acid in Patients With Moderately Severe Alcoholic Hepatitis (AH)
Acronym: TREAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Post-marketing reports of hepatotoxicity associated with obeticholic acid emerged in June 2017, investigators temporarily halted patient recruitment June 2017.
Sponsor: Naga P. Chalasani (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Naga P. Chalasani, Naga Chalasani, MD, FACG, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TREAT 002; 1U01AA021840-01 (NIH); U01AA021883 (NIH); U01AA021891 (NIH); U01AA021788 (NIH)
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 10 mg Obeticholic Acid (OCA) (Experimental): 10 mg Obeticholic Acid (OCA) Study medication will be administered orally, once daily for 6 weeks.
  Interventions: Drug: 10 mg Obeticholic Acid (OCA)

INTERVENTIONS:
Drug: Placebo — 1 tablet of placebo, taken orally daily with water, approximately 30 minutes prior to breakfast for 6 weeks.
  Arms: Placebo
Drug: 10 mg Obeticholic Acid (OCA) — 10 mg Obeticholic Acid (OCA) Study medication will be administered orally, once daily, approximately 30 minutes prior to breakfast for 6 weeks.
  Other Names: INT-747
  Arms: 10 mg Obeticholic Acid (OCA)

SUMMARY:
The main purpose of this study is to test the effectiveness of Obeticholic Acid when used in patients with moderately severe alcoholic hepatitis. The researchers suspect that individuals with alcoholic hepatitis have certain abnormalities in how their body handles bile acids (a product made by the liver on a daily basis) produced by the liver. Obeticholic acid has been shown to affect bile acid abnormalities and thus it is possible that obeticholic acid may improve liver condition in individuals with alcoholic hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 21 years with a diagnosis of acute AH. The diagnosis of acute alcoholic hepatitis will be based on clinical features and testing including hepatomegaly, jaundice, fever, leukocytosis, compatible liver biochemistries in the context of heavy alcohol consumption. A liver biopsy is not mandatory, but will be required to confirm the diagnosis if a firm diagnosis of AH cannot be made on clinical and laboratory criteria
* Moderate severity defined as MELD score > 11 and < 20
* Heavy alcohol consumption (defined as > 40 grams per day on average in women and > 60 grams per day on average in men for a minimum of 6 months and within the 6 weeks prior to study enrollment)
* Written informed consent
* Negative urine pregnancy test where appropriate
* Women of child bearing potential should be willing to practice contraception throughout the treatment period

Exclusion Criteria:

* Significant active infection (e.g., sepsis, or spontaneous bacterial peritonitis; SBP). Subjects can be reconsidered after the infection is under control.
* Serum creatinine > 2.5 mg/dL
* Must not be receiving systemic steroids > 1 week at the time of Screening or any experimental medicines for AH
* Presence of any other disease or condition that is interfering with the absorption, distribution, metabolism, or excretion of drugs including bile salt metabolism in the intestine. Patients who have undergone gastric bypass procedures will be excluded (gastric lap band is acceptable).
* Participation in another investigational drug, biologic, or medical device trial within 30 days prior to screening

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2018-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naga Chalasani, MD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - Indiana University, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Virgina Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Treatment
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Started | 11 | 8
Completed | 7 | 6
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 1 | 0
Period: Follow up
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Started | 7 | 6
Completed | 7 | 5
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA) | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.45 (9.61) | 50.375 (14.83) | 49.26 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 9 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: MELD Score Mean(SD)
Description: The Model for End-Stage Liver Disease (MELD) is a numerical scale, ranging from 6 (less ill) to 40 (gravely ill), used for liver transplant candidates age 12 and older. It gives each person a 'score' (number) based on how urgently he or she needs a liver transplant within the next three months.
Time Frame: Baseline to 6 weeks (Day 42)
Population: The decrease in MELD score from baseline to Day 42 was -3.4 in the OCA arm, and -2.2 in the placebo arm with an overall P-Value of 0.6170.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
units on a scale
  Baseline | 16.4 (2.2) | 14.9 (2.4)
  Day 42 | 13.9 (4.6) | 11.5 (6.8)
Statistical Analysis 1: Comparison: 10 mg Obeticholic Acid (OCA); Baseline; Test type: Superiority — The type of statistical test is superiority; p = 0.1758, t-test, 2 sided; Mean Difference (Net) = 1.5, Standard Deviation 2.4 — Two-sample t-test compared MELD score between OCA and placebo arms at baseline OCA arms had a mean (SD) of 14.9(2.4), Placebo arms had a mean (SD) of 16.4 (2.2)
Statistical Analysis 2: Comparison: 10 mg Obeticholic Acid (OCA); Day 42; Test type: Superiority — The type of statistical test is superiority; p = 0.3839, t-test, 2 sided; Mean Difference (Net) = 2.4, Standard Deviation 6.8 — Two-sample t-test compared MELD score between OCA and placebo arms at day 42 OCA arms had a mean (SD) of 11.5 (6.8), Placebo arms had a mean (SD) of 13.9(4.6)

2. Primary Outcome: Incidence of Serious Adverse Events (SAEs) During the Treatment Phase
Description: Number of subjects with one or more SAE are reported in relation to study medication (not related, unlikely, possible, probable, definite).
Time Frame: Baseline to 6 weeks (Day 42)
Population: Subjects with SAEs not related to OCA
Measure: Number; unit: Events
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
Events
  Not Related | 5 | 1
  Unlikely | 6 | 3
  Possible | 0 | 0
  Probable | 0 | 0
  Definite | 0 | 0

3. Primary Outcome: MELD Score Change From Baseline Mean(SD)
Description: as for outcome 1
Time Frame: Baseline to 6 weeks (Day 42)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
units on a scale | -2.2 (3.9) | -3.4 (5.9)

4. Secondary Outcome: Any SAEs During the Follow-up Phase
Description: as for outcome 2
Time Frame: Days 42 to 180
Measure: Number; unit: Events
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
Events
  Not Related | 5 | 5
  Unlikely | 3 | 1
  Possible | 0 | 0
  Probable | 0 | 0
  Definite | 0 | 0

5. Secondary Outcome: SAEs Attributable to the Study Medicine During the Treatment and Follow-up Phases
Description: as for outcome 2
Time Frame: Baseline to 180 days
Measure: Number; unit: Events
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
Events
  Not Related | 10 | 6
  Unlikely | 9 | 4
  Possible | 0 | 0
  Probable | 0 | 0
  Definite | 0 | 0

6. Secondary Outcome: Adverse Events (AEs) During the Treatment and Follow-up Phases
Description: Number of subjects with one or more AEs are reported in relation to study medication (not related, unlikely, possible, probable, definite).
Time Frame: Baseline to 180 days
Measure: Number; unit: Event
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
Event
  Not Related | 30 | 31
  Unlikely | 17 | 25
  Possible | 3 | 3
  Probable | 0 | 1
  Definite | 0 | 0

7. Secondary Outcome: Change in MELD Score at 90 and 180 Days
Description: as for outcome 1
Time Frame: Days 90 and 180
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
units on a scale
  Day 90 | -4.4 (2.8) | -6.0 (4.0)
  Day 180 | -4.0 (5.9) | -4.5 (2.3)

8. Secondary Outcome: Change in Child-Pugh Score at Day 42, 90 and 180 Days
Description: The Child-Pugh score is a system for assessing the prognosis - including the required strength of treatment and necessity of liver transplant - of chronic liver disease, primarily cirrhosis. It provides a forecast of the increasing severity of your liver disease and your expected survival rate. The Child-Pugh score is determined by scoring five clinical measures of liver disease. A score of 1, 2, or 3 is given to each measure, with 3 being the most severe. The total Child-Pugh range is 5-15, with 15 being the most severe.
Time Frame: Days 42, 90 and 180
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
units on a scale
  Day 42 | -1.6 (1.9) | -2.8 (1.7)
  Day 90 | -3.0 (1.2) | -3.0 (0.6)
  Day 180 | -2.3 (3.0) | -3.5 (0.8)

9. Secondary Outcome: Percentage of Participants Deceased at Day 42, 90 and 180
Description: Number of subjects deceased at day 42, 90, and 180.
Time Frame: Days 42, 90 and 180
Measure: Number; unit: percentage of mortality
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
percentage of mortality
  Day 42 | 9.09 | 0
  Day 90 | 9.09 | 0
  Day 180 | 9.09 | 0
Statistical Analysis 1: Comparison: Placebo; Day 42; Test type: Superiority — The type of statistical test is superiority; p = .3938, Log Rank; Survival Anaylsis = 0
Statistical Analysis 2: Comparison: 10 mg Obeticholic Acid (OCA); Day 90; Test type: Superiority — The type of statistical test is superiority; p = .3938, Log Rank; Survival Anaylsis = 0
Statistical Analysis 3: Comparison: 10 mg Obeticholic Acid (OCA); Day 180; Test type: Superiority — The type of statistical test is superiority; p = .3938, Log Rank; Survival Anaylsis = 0
Statistical Analysis 4: Comparison: Placebo; Day 42; Test type: Superiority — The type of statistical test is superiority; p = .3938, Log Rank; Survival Analysis = 0.09
Statistical Analysis 5: Comparison: Placebo; Day 90; Test type: Superiority — The type of statistical test is superiority; p = .3938, Log Rank; Survival Analysis = 0.09
Statistical Analysis 6: Comparison: Placebo; Day 180; Test type: Superiority — The type of statistical test is superiority; p = .3938, Log Rank; Survival Analysis = 0.09

10. Secondary Outcome: Rates of Hospitalization
Description: Number of subjects with one or more hospitalization are reported in relation to study medication (not related, unlikely, possible, probable, definite).
Time Frame: Baseline to 180 days
Measure: Number; unit: Events
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
Events
  Not Related | 4 | 6
  Unlikely | 0 | 0
  Possible | 0 | 0
  Probable | 0 | 0
  Definite | 0 | 0

11. Secondary Outcome: Changes in Intestinal Inflammation
Description: Early termination of the study resulted in insufficient numbers of participants in each arm to allow meaningful assessment of obeticholic acid effects on these secondary outcomes. Therefore these endpoints were not measured and no statistical analysis for these endpoints was done as they endpoints were not measured.
Time Frame: Baseline to Day 180
Population: Early termination of the study resulted in insufficient numbers of participants in each arm to allow meaningful assessment of obeticholic acid effects on these secondary outcomes. Therefore these endpoints were not measured and no statistical analysis for these endpoints was done as they endpoints were not measured.
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Changes in Serum Oxidative Stress.
Description: as for outcome 11
Time Frame: Baseline to 180 days
Population: as for outcome 11
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Length of Hospital Stays
Time Frame: Baseline to 180 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
Days | 1.9 (3.3) | 2.3 (2.5)
Statistical Analysis 1: Comparison: 10 mg Obeticholic Acid (OCA); Test type: Superiority — The type of statistical test is superiority; p = 0.8094, t-test, 2 sided; Mean Difference (Final Values) = .4, Standard Deviation 2.5

14. Secondary Outcome: Changes in Bacterial Translocation
Description: as for outcome 11
Time Frame: Baseline to 180 days
Population: as for outcome 11
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Changes in Cytokines
Description: as for outcome 11
Time Frame: Baseline to 180 days
Population: as for outcome 11
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Changes in Activation of Innate Immunity
Description: as for outcome 11
Time Frame: Baseline to 180 days
Population: as for outcome 11
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Discontinuation Rate During the Treatment and Follow-up Phases
Time Frame: Baseline to 180 days
Measure: Number; unit: Events
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 8
Events | 4 | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | 10 mg Obeticholic Acid (OCA)
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 5/11 | 6/8
Other Adverse Events (participants affected / at risk) | 9/11 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | 10 mg Obeticholic Acid (OCA) (N=8)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Blood electrolytes abnormal (Investigations) | 0 (0) | 1 (1)
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Kidney injury molecule-1 (Investigations) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | 10 mg Obeticholic Acid (OCA) (N=8)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Weigh Loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholestatic pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (5)
Electrocardiogram QT prolonged (Infections and infestations) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Faeces pale (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Jittery (General disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (3)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (4)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 4 (4) | 4 (5)
Penile swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Pulmonary physical examination abnormal (Investigations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Soft Tissue Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Varices oesophageal (Vascular disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT02039219/Prot_SAP_000.pdf